CLINICAL TRIAL: NCT02286440
Title: A Pharmacokinetic/Pharmacodynamic Genetic Variation Treatment Algorithm Versus Treatment As Usual for Adolescent Management Of Depression (Abbreviation Assurex AMOD)
Brief Title: A PK/PD Genetic Variation Treatment Algorithm Versus Treatment As Usual for Adolescent Management Of Depression
Acronym: AMOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul E. Croarkin, Paul E. Croarkin, D.O., M.S., Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14-005547
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Depression
Keywords: Depression; Genotyping; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GeneSight guided treatment (Experimental): GeneSight guided group will have their research psychiatrist make treatment recommendations based on test results
  Interventions: Other: AssureRx GeneSight genotyping results
- Treatment as usual group (Active Comparator): Treatment as usual group will have treatment recommendations based on clinical judgment
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: AssureRx GeneSight genotyping results
  Arms: GeneSight guided treatment
Other: Treatment as usual
  Arms: Treatment as usual group

SUMMARY:
The overall goal of this investigator-initiated trial is to evaluate the impact of platform algorithm products designed to rapidly identify pharmacokinetic (PK) and/or pharmacodynamic (PD) genomic variation on treatment outcome of depression in adolescents. This new technology may have the potential to optimize treatment selection by improving response, minimizing unfavorable adverse events / side effects and increasing treatment adherence

DETAILED DESCRIPTION:
Treatment seeking adolescent patients with a moderate to severe major depressive episode defined as a 40 or greater on Childhood Depression Rating Scale-Revised (CDRS-R) will be invited to participate in this study evaluating the GeneSight® platform. This new technology can rapidly assess PK and PD genetic variation that can potentially impact antidepressant, anti-psychotic, and stimulant treatment selection. These patients will have GeneSight® testing and will be randomized to one of two groups. In Group 1 (n=138), GeneSight® testing results will be available to the patient's treating clinician prior to treatment selection. In Group 2 (n=138), testing results will not be available to the patient's research treating clinician. However, all testing results will be made available to all participants and clinicians after the 8-week trial (upon completion of blinded assessments at week 8). The patients and the clinical raters will be blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-18, male or female, any race/ethnicity
* Treating clinician, patient, and family feel that pharmacotherapy is indicated as part of a comprehensive treatment plan.
* Major depressive episode diagnosis or bipolar disorder based on KSADS-PL semi-structured psychiatric interview with a severity criteria-40 or greater on Childhood Depression Rating Scale-Revised (CDRS-R)
* Ability to provide informed consent

Exclusion Criteria:

* Inability to speak English
* Inability or lack of willingness to provide informed consent and assent.
* Axis I diagnoses: Autism Spectrum Disorder, Anorexia Nervosa, Schizophreniform, and Schizophrenia.
* Psychotropic medication change (including dosage) between screening & randomization visits.
* Patients who meet DSM 5 criteria for any significant current substance use disorder other than nicotine, caffeine, or cannabis. Must have at least early, partial or full, remission X 3 months
* Serious suicidal risk and/or in need of immediate hospitalization as judged by the investigator.
* Significant unstable medical condition.
* Anticipated inability to attend scheduled study visits.
* Patients who in the judgment of the Investigator may be unreliable or uncooperative with the evaluation procedure outlined in this protocol.
* Cytochrome (CYP) & serotonin transporter genomic testing within 5 years.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 179 (Actual)
Dates: Start 2015-02; Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Baseline to endpoint change in depression | 8 weeks
  The primary outcome measure is the baseline to endpoint change in the Children's Depression Rating Scale, Revised (CDRS-R).

SECONDARY OUTCOMES:
Improvement of depressive symptoms | 8 weeks
  Quick Inventory of Depressive Symptomatology Adolescent Clinician Rated Form (QIDS-A17 CR)
Improvement of depressive symptoms | 8 weeks
  Quick Inventory of Depressive Symptomatology Adolescent Self-Report (QIDS-A17 SR)
Improvement of depressive symptoms | 8 weeks
  Quick Inventory of Depressive Symptomatology Adolescent Self-Report - Parent [(QIDS-A17 SR (P)
Improvement of depressive symptoms | 8 weeks
  Clinical Global Impression (CGI) scale
Improvement of depressive symptoms | 8 weeks
  Global Assessment Scale (CGAS)
Improvement of depressive symptoms | 8 weeks
  General Behavior Inventory Parent Version (P-GBI) (subscales mania and sleep) Short Form
Improvement of depressive symptoms | 8 weeks
  Treatment adherence based on concordance vs. non-concordance of gene test results and clinical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paul Croarkin, D.O., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nooraeen S, Croarkin PE, Geske JR, Shekunov J, Orth SS, Romanowicz M, Frye MA, Vande Voort JL. High Probability of Gene-Drug Interactions Associated with Medication Side Effects in Adolescent Depression: Results from a Randomized Controlled Trial of Pharmacogenetic Testing. J Child Adolesc Psychopharmacol. 2024 Feb;34(1):28-33. doi: 10.1089/cap.2023.0043. PMID 38377526
- [Derived] Vande Voort JL, Orth SS, Shekunov J, Romanowicz M, Geske JR, Ward JA, Leibman NI, Frye MA, Croarkin PE. A Randomized Controlled Trial of Combinatorial Pharmacogenetics Testing in Adolescent Depression. J Am Acad Child Adolesc Psychiatry. 2022 Jan;61(1):46-55. doi: 10.1016/j.jaac.2021.03.011. Epub 2021 Jun 5. PMID 34099307
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials